CLINICAL TRIAL: NCT05064007
Title: The Power of Sound and Music Interventions for Older Adults With Mild Cognitive Impairment
Brief Title: Sound and Music for Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00295386; R21AG078917 (NIH)
Record Dates: First submitted 2021-09-21; First posted 2021-10-01 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): this group will be exposed to condition A first, then B, and C
  Interventions: Behavioral: A: 40 Hz music; Behavioral: B: 40 Hz sound; Behavioral: C: Preferred music
- 2 (Experimental): this group will be exposed to condition B first, then C, and A
  Interventions: Behavioral: A: 40 Hz music; Behavioral: B: 40 Hz sound; Behavioral: C: Preferred music
- 3 (Experimental): this group will be exposed to condition C first, then A, and B
  Interventions: Behavioral: A: 40 Hz music; Behavioral: B: 40 Hz sound; Behavioral: C: Preferred music

INTERVENTIONS:
Behavioral: A: 40 Hz music — The participant will listen to the 40 Hz music playlist one hour each day, 5 days a week for 4 weeks
Behavioral: B: 40 Hz sound — The participant will listen to the 40 Hz sound playlist one hour each day, 5 days a week for 4 weeks
Behavioral: C: Preferred music — The participant will listen to the preferred music playlist one hour each day, 5 days a week for 4 weeks

SUMMARY:
Emerging studies in humans found that 40 Hz sound induces neural gamma oscillation and enhanced cognitive function in older adults with and without Alzheimer's Disease. We will compare a 40 Hz music intervention to both 40 Hz sound and music alone in a clinical cohort of older adults with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling
2. amnesia mild cognitive impairment
3. Preserved function
4. No dementia

Exclusion Criteria:

1. known diagnosis of schizophrenia or Parkinson's disease;
2. severe hearing impairment;
3. presence of an acute medical or psychiatric condition which would interfere with the subject's ability to follow the study protocol realistically

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2025-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JUNXIN LI, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from multiple sources including community recruitment, memory clinics, and online recruitment platforms.
Pre-assignment Details: A total of 52 participants were consented. Fifteen participants who withdrew while waiting for randomization or 1st treatment were excluded. 37 participants were randomized.
Groups:
- Sequence 1: This Group Will be Exposed to Condition A First, Then B, and C; Sequence 2: This Group Will be Exposed to Condition B First, Then C, and A; Sequence 3: This Group Will be Exposed to Condition C First, Then A, and B: A: 40 Hz music: The participant will listen to the 40 Hz music playlist one hour each day, 5 days a week for 4 weeks
  B: 40 Hz sound: The participant will listen to the 40 Hz sound playlist one hour each day, 5 days a week for 4 weeks
  C: Preferred music: The participant will listen to the preferred music playlist one hour each day, 5 days a week for 4 weeks
Period: First Intervention (4 Weeks)
Arm/Group | Sequence 1: This Group Will be Exposed to Condition A First, Then B, and C | Sequence 2: This Group Will be Exposed to Condition B First, Then C, and A | Sequence 3: This Group Will be Exposed to Condition C First, Then A, and B
Started | 14 | 10 | 13
Completed | 14 | 10 | 12
Not Completed | 0 | 0 | 1
Period: Washout (10-14 Days)
Arm/Group | Sequence 1: This Group Will be Exposed to Condition A First, Then B, and C | Sequence 2: This Group Will be Exposed to Condition B First, Then C, and A | Sequence 3: This Group Will be Exposed to Condition C First, Then A, and B
Started | 14 | 10 | 12
Completed | 12 | 10 | 10
Not Completed | 2 | 0 | 2
Period: Second Intervention (4 Weeks)
Arm/Group | Sequence 1: This Group Will be Exposed to Condition A First, Then B, and C | Sequence 2: This Group Will be Exposed to Condition B First, Then C, and A | Sequence 3: This Group Will be Exposed to Condition C First, Then A, and B
Started | 12 | 10 | 10
Completed | 11 | 10 | 10
Not Completed | 1 | 0 | 0
Period: Washout (10-14 Days)
Arm/Group | Sequence 1: This Group Will be Exposed to Condition A First, Then B, and C | Sequence 2: This Group Will be Exposed to Condition B First, Then C, and A | Sequence 3: This Group Will be Exposed to Condition C First, Then A, and B
Started | 11 | 10 | 10
Completed | 9 | 10 | 8
Not Completed | 2 | 0 | 2
Period: Third Intervention (4 Weeks)
Arm/Group | Sequence 1: This Group Will be Exposed to Condition A First, Then B, and C | Sequence 2: This Group Will be Exposed to Condition B First, Then C, and A | Sequence 3: This Group Will be Exposed to Condition C First, Then A, and B
Started | 9 | 10 | 8
Completed | 8 | 9 | 8
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence ABC: this group will be exposed to condition A first, then B, and C
  A: 40 Hz music: The participant will listen to the 40 Hz music playlist one hour each day, 5 days a week for 4 weeks
  B: 40 Hz sound: The participant will listen to the 40 Hz sound playlist one hour each day, 5 days a week for 4 weeks
  C: Preferred music: The participant will listen to the preferred music playlist one hour each day, 5 days a week for 4 weeks
- Sequence BCA: this group will be exposed to condition B first, then C, and A
  A: 40 Hz music: The participant will listen to the 40 Hz music playlist one hour each day, 5 days a week for 4 weeks
  B: 40 Hz sound: The participant will listen to the 40 Hz sound playlist one hour each day, 5 days a week for 4 weeks
  C: Preferred music: The participant will listen to the preferred music playlist one hour each day, 5 days a week for 4 weeks
- Sequence CAB: This group will be exposed to condition C first, then A, and B
  A: 40 Hz music: The participant will listen to the 40 Hz music playlist one hour each day, 5 days a week for 4 weeks
  B: 40 Hz sound: The participant will listen to the 40 Hz sound playlist one hour each day, 5 days a week for 4 weeks
  C: Preferred music: The participant will listen to the preferred music playlist one hour each day, 5 days a week for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB | Total
Number analyzed (Participants) | 14 | 10 | 13 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (7.8) | 68.7 (6.3) | 66.7 (7.1) | 67.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 6 | 23
  Male | 6 | 1 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 6 | 8 | 23
  White | 4 | 3 | 5 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Episodic Memory Assessed by the Cogstate Alzheimer's Battery
Description: The composite episodic memory score is calculated as a Z-score, representing the sum of the Z-scores across three Cogstate computerized assessments: One Card Learning, International Shopping List, and Delayed Recall. For each test, a Z-score is calculated relative to the first baseline assessment of all included subjects, using the formula (score - mean at first baseline assessment) / standard deviation at first baseline assessment. The composite Z-score is then calculated by summing these individual Z-scores. A composite Z-score of 0 corresponds to performance exactly at the study-sample mean at the first baseline assessment. Positive, or higher, composite Z-scores reflect better episodic-memory performance-they show how many standard deviations above the baseline mean the summed score lies. Conversely, negative, or lower, composite Z-scores reflect poorer episodic-memory performance, indicating how many standard deviations below the baseline mean the score falls.
Time Frame: Baseline and 4 weeks
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: z score
Groups:
- 40 Hz Music: Participants who were assigned to listen to the 40 Hz music playlist one hour each day, 5 days a week, for 4 weeks
- 40 Hz Sound: The participants were assigned to listen to the 40 Hz sound playlist one hour each day, 5 days a week for 4 weeks
- Preferred Music: The participants who were assigned to listen to the preferred music playlist one hour each day, 5 days a week for 4 weeks
Arm/Group | 40 Hz Music | 40 Hz Sound | Preferred Music
Number analyzed (Participants) | 33 | 28 | 30
z score
  Baseline | -0.0746 (2.5595) | 0.0700 (2.37813) | 0.0593 (2.1298)
  Post-intervention | 0.5137 (2.57731) | 0.553 (2.50150) | 0.1614 (2.34475)

2. Primary Outcome: Global Cognition Assessed by the Cogstate Alzheimer's Battery
Description: The composite global cognitive score is expressed as a Z-score obtained by summing the Z-scores from six Cogstate computerized assessments: Identification, Detection, One Card Learning, One Back, International Shopping List-Delayed Recall, and Groton Maze Learning. For each task, an individual Z-score is calculated with reference to the first baseline assessment of all enrolled participants using the formula (individual score - baseline mean) / baseline standard deviation. These task-specific Z-scores are then summed to yield the composite value. A composite Z-score of 0 denotes performance exactly at the study-sample mean at the first baseline assessment. Positive-or higher-composite Z-scores reflect better global cognitive performance because they indicate performance a given number of standard deviations above that first baseline mean, whereas negative-or lower-composite Z-scores reflect poorer performance by indicating the number of standard deviations below the mean.
Time Frame: Baseline and Immediate after 4-week intervention
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | 40 Hz Music | 40 Hz Sound | Preferred Music
Number analyzed (Participants) | 30 | 29 | 25
z score
  Baseline | 8.3831 (35.542) | 5.5993 (28.40206) | 15.3345 (27.42554)
  Post-intervention | 18.6907 (28.38671) | 16.2249 (28.2289) | 10.4428 (29.44993)

ADVERSE EVENTS:
Time Frame: During study participation, approximately 18 weeks
Groups:
- 40 Hz Music; Preferred Music: No adverse events were reported
- 40 Hz Sound: Three participants reported hearing buzzing sounds lasting 5 to 15 minutes following the completion of the listening sessions
Arm/Group | 40 Hz Music | 40 Hz Sound | Preferred Music
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/34 | 0/30 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT05064007/Prot_SAP_000.pdf